CLINICAL TRIAL: NCT06870864
Title: Role of Conservative Management in Adhesive Intestinal Obstruction Versus Operative Management
Brief Title: Conservative Versus Operative Management in Adhesive Intestinal Obstruction
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Osama Khaled Ahmed, Principal investigator, Sohag University
Other Study IDs: Soh-Med--25-1-09MS
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Adhesive Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the role of Conservative management in patients with adhesive Intestinal Obstruction Regarding the selection criteria of the patients, duration of conservative route, success rate, and recurrence of adhesions and avoiding the surgical route complications.

DETAILED DESCRIPTION:
Adhesive Intestinal Obstruction is very common and represents a serious life threatening condition, which can be caused by congenital band, following abdominal surgeries and other medical conditions like tuberculosis.

The management options for adhesive intestinal obstruction (AIO) could be operative treatment (open-laparoscopy) or non-operative (conservative management) according to many reasons.

Some reports indicate that the operative management for adhesive Intestinal obstruction lead to further adhesions in the future in addition to other possible complications (anaesthetic - iatrogenic injury during adhesolysis - wound site infections - illius-long hospital stay).

The Conservative route is recommended in all patients except those with signs of peritonitis, strangulation, or bowel ischemia which would have been diagnosed during physical examination and imaging.

A few studies compared the advantages, safety, and less complications of Conservative versus operative management. Therefore, this study will be conducted on patients with adhesive Intestinal Obstruction to compare the effectiveness of Conservative versus operative management regarding the selection criteria for the patients, the duration of the Conservative route, things to be done and what need to be observed during the conversation time.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-70 years.
* Both sexes.
* Complete \ Partial adhesive Intestinal Obstruction, with CT Abdomen and pelvis with oral and IV Contrast.

Exclusion Criteria:

* Patients with signs of Strangulation
* Patients with signs of peritonitis.
* Patients with signs of bowel ischemia
* Failure of Conservative management for more than 72 hours.
* Vitally unstable patients
* Patients with comorbidities which need rapid interventions.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with adhesive Intestinal Obstruction at Department of General Surgery, Oncological and Laparoscopic Surgeries, Sohag University Hospitals, Sohag, Egypt
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
X-Ray Changes | 72 Hours
  Daily Chest Abdomen X-ray Erect copies to evaluate the improvement of the Intestinal Obstruction through evaluation of the X-ray findings (Air fluid levels).
Passability Status | 72 Hours
  Daily history taking records and per rectal examination findings to evaluate the passability status (stool /flatus)
Hospital Stay Duration | from 3 to 5 days.
  The Conservative management in patients with adhesive Intestinal Obstruction will avoid them the surgical route which requires long hospital stay postoperative
Vomiting | 72 Hours
  Frequency and severity of vomiting will be collected to help in prognosis prediction
Abdominal Signs | 72 Hours
  Data collected about Daily abdominal examination findings (Distention, Intestinal sounds, abdominal pain and Per rectal examination).

SECONDARY OUTCOMES:
Recurrence of Attacks | two years previous the onset of the current attack. (During the last two years before the admission)
  past history about the previous attacks of the adhesive Intestinal Obstruction
Past Surgical History | two years previous the onset of the current attack. (During the last two years before the admission)
  Detailed history about the previous operations to determine the relationship between different operations and adhesive Intestinal Obstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt